CLINICAL TRIAL: NCT03542942
Title: Exclusion of Non-involved Uterus Form the Target Volume: an Individualized Treatment for Locally Advanced Cervical Cancer Using Modern Radiotherapy and Imaging Techniques
Brief Title: Exclusion of Non-involved Uterus From the Target Volume in Locally Advanced Cervical Cancer
Acronym: EXIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B670201526181
Record Dates: First submitted 2018-05-03; First posted 2018-05-31 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Uterine Cervical Neoplasms
Keywords: locally advanced; radiotherapy; DW-MRI; target volume
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment with EXIT-target volume (Other): The radiotherapeutic treatment plan is based on an EXIT-target volume in which the non-involved uterus is excluded from the target volume. All other delineations are performed conform standard of care.
  Interventions: Other: treatment with EXIT-target volume

INTERVENTIONS:
Other: treatment with EXIT-target volume — exclusion of the unaffected part of the uterus out of the treatment field

SUMMARY:
Both toxicity and local relapse are major concerns in the treatment of locally advanced cervical cancer. The purpose of this study is to ameliorate both by integrating modern imaging (diffusion weighted magnetic resonance imaging; DW-MRI) into the treatment planning of modern radiotherapy. We want to evaluate the safety and effect of excluding the unaffected uterus (as determined on magnetic resonance imaging) from the treatment field. Meanwhile we want to explore the possible use of apparent diffusion coefficient values (DW-MRI) as biomarker of treatment response.

DETAILED DESCRIPTION:
In our previous research we successfully implemented Intensity Modulate Arc Therapy with concurrent administration of cisplatin 40mg/m2 weekly (IMAT-C) in the multimodality treatment of Locally Advanced Cervical Cancer (LACC) . By delivering a higher biological dose to the tumor and lowering the dose to the Organs at Risk (OARs), toxicity significantly dropped and local control improved. However, there remains room for improvement for both toxicity and response to the treatment. Macroscopic tumor rest on hysterectomy reflects the existence of chemoradiation (CRT) resistant foci and correlates with outcome. We hypothesize that both radiotherapy (RT)-related toxicity (a) as well as local response on CRT (b) can be improved by respectively:

1. Reducing the dose on OARs by omitting iconographical non tumor-bearing parts of the uterus from the Clinical Target Volume (CTV).
2. Performing a dose-escalation to those regions within the gross target volume (GTV) pointed out by Diffusion Weighted Magnetic Resonance Imaging (DW-MRI) to be at risk for treatment failure.

To objectivize our hypotheses, we aim at:

1. Demonstrating that omitting iconographical unaffected uterus from the treatment volume leaves no tumor behind in the non-targeted parts of the uterus, leads to lower doses to the OARs and decreases (acute) toxicity.
2. Validating that a high baseline apparent diffusion coefficient (ADC) and an increase in ADC 2 weeks after start of CRT, for the whole tumor as well as for intra-tumoral regions, is prognostic for residual tumor on hysterectomy specimen and to consider the possibility for a further dose-escalation on tumors/intratumoral regions at risk for treatment failure.

Importance to the field: Both toxicity and local relapse are major concerns in the treatment of LACC. Grade ≥ 2 toxicity influences daily life of patients significantly and is present in the majority of patients treated and even with image guided BT local relapse remains the major cause of treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven carcinoma of the uterine cervix
* locally advanced disease (FIGO IB2 or >FIGO IIB or node positive) proven by clinical examination, 18-fluorodeoxyglucose positron emission tomography scan (18FDG PET-CT) and MRI
* no more than 2 distant metastases (other than para-aortic lymph nodes);
* WHO 0-2;
* adequate kidney function for CRT, if inadequate kidney function radiotherapy can be the sole therapeutic regimen;
* not pregnant or breastfeeding
* absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; - willing and able to sign a written informed consent.

Exclusion Criteria:

* Patients unable to undergo MRI for any reason.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
safety: abscence of tumor in the non-involved and non-high doses irradiated part of the uterus | within 3 months after last inclusion
  abscence of tumor in the non-involved (as determined on the pre-treatment MRI) and non-high doses irradiated part of the uterus in the hysterectomy specimen after CRT

SECONDARY OUTCOMES:
dosimetry | within 3 months after last inclusion
  dosimetric comparison of dose on the OARs when comparing study treatment plans compared to treatment of the whole uterus at high doses
number of participants with treatment-related adverse events as assessed by the radiotherapy oncology group toxicity criteria and CTCAEv4.0 for hematology | during treatment. 10 days, 1 months and 3 months after ending treatment
  evaluation of acute toxicity, grade 0 (no toxicity) to grade 5 (treatment related death).
number of participants with treatment-related adverse events as assessed by the radiotherapy oncology group toxicity criteria and CTCAEv4.0 | 6, 12, 18 and 24 months after treatment.
  evaluation chronic toxicity, grade 0 (no toxicity) to grade 5 (treatment related death).
local, regional and distant control | 1, 3, 6, 12,18 and 24 months after treatment
  defined as absence of disease at the primary tumor bed, the regional lymph nodes and distant sites
Correlation of high-Risk regions on IMaging (DW-MRI) with Pathology and regression pattern analysis (CRIMP). | Within 6 months after surgery of the last patient
  The MRI at fixed time points will be supplemented with diffusion weighing (DW). The ultimate aim is the correlation of tumoral ADC-values of the different DW-MRI with the pathology in order to predict therapy resistance or response to CRT at an early stage or even before start.

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Vandecasteele, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Radiotherapy Department Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be shared. Decision is made upon request.

REFERENCES:
- [Derived] Vandecasteele K, Tummers P, Van Bockstal M, De Visschere P, Vercauteren T, De Gersem W, Denys H, Naert E, Makar A, De Neve W. EXclusion of non-Involved uterus from the Target Volume (EXIT-trial): an individualized treatment for locally advanced cervical cancer using modern radiotherapy and imaging techniques. BMC Cancer. 2018 Sep 17;18(1):898. doi: 10.1186/s12885-018-4800-0. PMID 30223802